CLINICAL TRIAL: NCT02255773
Title: Exploring the Neuro-Immune Basis of Cancer-Related Fatigue Using Behavioral Measures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014-0511; NCI-2015-00012 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2014-09-26; First posted 2014-10-03 (Estimated); Last update posted 2024-03-29 (Actual); Status verified 2024-03

CONDITIONS: Head and Neck Cancer
Keywords: Head and Neck Cancer; HNC; Moderate to severe fatigue; Computerized tasks; Questionnaires; Surveys; Disease-free adult males; Cancer survivors
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- High-Fatigue Head and Neck (HNC) Cancer Survivors (Other): Participants undergo assessment with three validated computerized tasks designed to measure the neurobehavioral domains of interest: the Effort Expenditure for Rewards Task (EEfRT), an associative learning task, and a set-switch task. Participants complete questionnaires assessing mood, somatic symptoms, and sleep quality, including the Multidimensional Fatigue Symptom Inventory-Short Form (MFSI-SF), the Checklist Individual Strength (CIS), and others. A 10-mL blood sample drawn for assessment of inflammatory markers and COMT and DAT1 genotype.
  Interventions: Behavioral: Computerized Tasks; Behavioral: Questionnaires
- Low-Fatigue Head and Neck (HNC) Cancer Survivors (Other): Participants undergo assessment with three validated computerized tasks designed to measure the neurobehavioral domains of interest: the Effort Expenditure for Rewards Task (EEfRT), an associative learning task, and a set-switch task. Participants complete questionnaires assessing mood, somatic symptoms, and sleep quality, including the Multidimensional Fatigue Symptom Inventory-Short Form (MFSI-SF), the Checklist Individual Strength (CIS), and others. A 10-mL blood sample drawn for assessment of inflammatory markers and COMT and DAT1 genotype.
  Interventions: Behavioral: Computerized Tasks; Behavioral: Questionnaires

INTERVENTIONS:
Behavioral: Computerized Tasks — 3 computerized tasks completed to assess motivation, learning of goal-directed and habitual behavior, and flexibility in switching between behavior strategies. It should take about 60 minutes to complete all three tasks.
Behavioral: Questionnaires — Completion of 8 questionnaires about mood, fatigue, sleep quality, and other symptoms. It should take about 30 minutes to complete these questionnaires.
  Other Names: Surveys

SUMMARY:
The goal of this research study is to learn more about fatigue and how it affects your behavior as well as your willingness to learn new behaviors.

DETAILED DESCRIPTION:
If you agree to take part in this study, the following tests and procedures will be performed:

* Blood (about 3 teaspoons) will be drawn to test for markers of inflammation and to test for genes related to brain signaling. Markers of inflammation are found in the blood and may be related to your fatigue and other symptoms.
* You will complete three tasks on a computer. Some of the tasks are easy and you are already used to them, but other ones will require some learning. You will be given written instructions on how to complete them. The tasks will be completed in or near the Head and Neck Cancer outpatient clinics. It should take about 60 minutes to complete all three tasks.
* You will complete 9 questionnaires about your mood, fatigue, sleep quality, and other symptoms. It should take about 30 minutes to complete these questionnaires.

The questionnaires will be given a code number and stored in a locked file cabinet at MD Anderson. No identifying information will be directly linked to your questionnaires. Only the researcher in charge of the study will have access to the code numbers and be able to link the questionnaires to you.

Length of Study:

After you have completed the blood draw, the computerized tasks, and the questionnaires, your participation on this study will be over.

Additional Information:

Any information about your symptoms that is collected as part of this study is for research purposes only. The questionnaires will only be used for the purposes of this study and will be destroyed after the study results have been reported.

If you describe a symptom as being severe on the symptom questionnaire, a study staff member will ask you if you have already told or plan to tell your doctor or nurse about the symptom. If you have not already told your doctor or nurse, a study staff member will tell your doctor or nurse about the symptom for you.

This is an investigational study.

Up to 60 participants will be enrolled in this study. All will take part at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Male patients at least 18 years old.
2. Patients who completed either definitive or postoperative radiation or chemoradiation therapy for head and neck cancer within the past 6 weeks to 120 months.
3. Patients who speak English.
4. Patients who are willing and able to review, understand, and provide written consent.
5. Patients who agree to comply with all study procedures.

Exclusion Criteria:

1. Patients with clinical evidence of active persistent cancer or progressive disease after completing planned cancer therapy, or with active recurrent cancer.
2. Patients with potential medical or other underlying causes of fatigue, as determined by the treating physician or Principal Investigator.
3. Patients with underlying cardiac or pulmonary disease resulting in dyspnea, hypoxia, or hypercapnia.
4. Patients with major depressive disorder or severe depression (a score of 22 or greater on the Center for Epidemiologic Studies Depression (CES-D)); for scores of 16 or higher, we will notify the patient's treating physician within 1 working day of the screening to allow for appropriate management or referral.
5. Patients currently taking, or having taken within the previous 1 month, armodafinil, modafinil, amphetamine, or methylphenidate.
6. Patients who are enrolled and receiving active treatment in a symptom intervention trial or who are in the treatment phase of a clinical trial.
7. Patients experiencing moderate to severe pain (4 or higher on a 0 to 10 scale) at the time of screening.
8. Patients who cannot distinguish between the red and blue stimuli of the set-switch task.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2014-11-04 (Actual); Primary Completion 2024-03-27 (Actual); Study Completion 2024-03-27 (Actual)

PRIMARY OUTCOMES:
Fatigue Comparison in Male Head and Neck Cancer Survivors | 1 day
  Endpoint for Effort Expenditure for Rewards Task (EEfRT) is ratio of hard task choices (number of hard task choices/total choices) across levels of probability. Endpoints for associative learning task are number of trials until reaching the a priori defined learning criterion (three consecutive correct responses for each association), indicating goal-directed learning, and number of trials between reaching this criterion and reaching asymptote in the reaction times, indicating establishment of habitual behavior. Set-switching task primary endpoints is difference in reaction times and number of errors between "no-switch" and "switch" trials.

SECONDARY OUTCOMES:
Markers of Inflammation and Fatigue | 1 day
  Frequency of each COMT genotype (Val/Val; Met/Met; Val/Met) compared between high-fatigue and low-fatigue survivors.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Dantzer, DMV,PHD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org